CLINICAL TRIAL: NCT04719806
Title: Textural Analysis in Low Grade Gliomas on Pre Operative MRI Exams to Determine Molecular Status : a Retrospective Study
Brief Title: MR Textural Analysis in Low Grade Gliomas
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 20radio01
Record Dates: First submitted 2021-01-18; First posted 2021-01-22 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-01

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — brain tumor surgically removed or biopsied
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
WHO classification of low grade gliomas now relies on tumoral molecular patterns, especially on IDH mutation and 1p/19q co deletion status. Textural analysis on medical imaging is studied in several fields, and could provide help in patients with brain tumor due to possible complications of brain biopsy. The purpose of this study is to determine if specific textural signature on MR imaging could be found for low grade gliomas. The investigators included patients with LGG diagnosed at CHU of Nice abd whose first MRI was available on the PACS of the CHU. Textural data are extraxted by tumoral contouring and specific logiciel (LifeX) and histopathologic data are assessed for each patient. Then the investigators analyze it to dtermine if textural indices can predict molecar status.

ELIGIBILITY:
Inclusion Criteria:

LGG diagnosed at CHU of Nice abd whose first MRI was available on the PACS of the CHU

Exclusion Criteria:

-

Ages: 19 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lower grade gliomas diagnosed at CHU of Nice with pre operative MRI and molecular data available
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
review of MRI images to find clues that can predict molecular status | 9 years

CONTACTS AND LOCATIONS:
Locations (1):
- Nice University Hospital, Nice, France

IPD SHARING:
Plan to Share IPD: No